CLINICAL TRIAL: NCT05509582
Title: Extension Study (Extended Access) of Syk-inhibition Using Fostamatinib to Treat Post-Transplant Immune-mediated Cytopenias
Brief Title: Extension Study (Extended Access) of Syk-inhibition Using Fostamatinib to Treat Posttransplant Immune-mediated Cytopenias
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No responders in parent protocol 000758; this follow-on protocol not activated and PI leaving NIH
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10000760; 000760-H
Record Dates: First submitted 2022-08-19; First posted 2022-08-22 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Immune Mediated Anemia; Immune Mediated Thrombocytopenia; Chronic GVHD
Keywords: Allogeneic Hematopoietic Stem Cell Transplant; Graft Versus Host Disease; Spleen Tyrosine Kinase (Syk) Inhibitor
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Bronchiolitis Obliterans Syndrome; Graft vs Host Disease | interventions — fostamatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Fostamatinib Arm (Experimental): The subjects will receive oral fostamatinib daily for up to 2 years.
  Interventions: Drug: fostamatinib

INTERVENTIONS:
Drug: fostamatinib — Subjects will receive fostamatinib at the same dose as the dose they receive at the time of rollover. The dose could be reduced to 100mg daily, 150 mg daily, 100 mg twice a day if a dose-limiting adverse event occurred. After the initial 12 weeks on the extended access (total of 24 weeks of treatment), subjects will have the option to start tapering fostamatinib if they are maintaining hematologic recovery. Subjects with persistent (=2 readings, 2 weeks apart) loss of hematologic response, defined as Hb<9g/dL and/or PLT< 30 X 10^9/L can increase their dose to next higher dose. Once count stabilization again occurs, a slow dose reduction to next lowest dose (100mg or 150mg) can be performed to identify the lowest dose necessary to keep counts over these thresholds.

SUMMARY:
Background:

People who have a blood stem cell transplant can sometimes develop cytopenia. This means that their levels of one or more types of blood cell, such as the red cells or platelets, are lower than they should be. This can occur because a person s immune system might attack these cells after a stem cell transplant. Up to 20% of people who have blood stem cell transplants develop cytopenias, which can lead to anemia, severe bleeding, infections, and other problems. Treatments are needed to help keep blood cell levels stable after blood stem cell transplant.

Objective:

To evaluate the long-term effects of a study drug (fostamatinib) in people with cytopenia after a blood stem cell transplant.

Eligibility:

People who responded well to fostamatinib in an earlier study.

Design:

Participants will be screened. They will have a physical exam and blood tests.

Fostamatinib is an oral tablet taken by mouth. Participants will take the pills at the same dose and frequency as they did during the previous study. They will take the pills for up to 21 months. The dosage of the drug may be reduced over time if their blood cell levels are stable.

Participants will have a medical assessment every month. This can be with their local doctor or at the NIH clinic.

Participants will have blood tests every 3 months.

Participants will have a follow-up visit after they stop taking the drug. Their vital signs will be taken, and they will have blood drawn. They will answer questions about their health.

DETAILED DESCRIPTION:
Study Description:

This is an extension trial of a phase II study which is designed to evaluate the long-term safety and efficacy of fostamatinib in the treatment of post-transplant cytopenias as assessed by hematologic improvement in anemia and/or thrombocytopenia following an additional 12-84 weeks of treatment on the initial phase II trial. The subjects who are deemed responders to the initial 12-week treatment, will be candidates to enroll onto the extension trial for up to 2 years of treatment.

Objectives:

The primary objective is to evaluate the efficacy for the use of fostamatinib in subjects with post-transplant anemia and/or thrombocytopenia at the end of total 24 weeks of treatment.

The secondary objectives are to evaluate the long-term efficacy of subjects on fostamatinib while weaning off fostamatinib treatment either partially or completely.

Endpoints:

The primary endpoint is:

-Proportion of subjects who are able to maintain hematologic recovery (as defined below) by the end of 12 weeks on the extended access trial (total of 24 weeks fostamatinib treatment).

Hematologic recovery is defined as:

-Hemoglobin >= 10 g/dL (or at least >= 2 g/dL above baseline) in subjects enrolled with posttransplant anemia. In subjects with symptomatic anemia, a hemoglobin increase of at least >= 2 g/dL above baseline is required

OR

-Platelets >= 50 X 10^9/L (or at least >= 20 X 10^9/L above baseline) in subjects enrolled with posttransplant thrombocytopenia

OR

-Both of the above criteria in subjects with posttransplant Evans syndrome

The secondary endpoints:

* Proportion of subjects who are able to taper off fostamatinib by >33% while maintaining hematologic recovery as outlined above at the end of the treatment.
* Proportion of subjects who are able to completely taper off fostamatinib while maintaining hematologic recovery as outlined above at the end of the treatment.
* Change in corticosteroid dose in the total 24 weeks on fostamatinib, measured by median daily weight-based prednisone-equivalent corticosteroid dose in a week, from week 1 to week 24
* Change in the dose of other immunosuppressive agents in the total 24 weeks on fostamatinib, measured by median daily dose of the immunosuppressant in a week, from week 1 to week 24

ELIGIBILITY:
* INCLUSION CRITERIA:
* Subjects who were enrolled on phase II trial of fostamatinib and deemed responders at the time of rollover to the extended access trial which is defined as:

  * Hemoglobin >= 9 g/dL (or at least >= 1 g/dL above baseline) in subjects enrolled with posttransplant anemia without transfusion support, at least once during the 12-week phase II trial.

OR

--Platelets >= 30 X 10^9/L (or at least >= 10 X 10^9/L above baseline) without transfusion support, at least once during the 12-week phase II trial, in subjects enrolled with posttransplant thrombocytopenia

OR

--Either of the above criteria in subjects with posttransplant Evans syndrome

* Completed the end of study visit (week 12) on the initial protocol (A Phase II Study of Syk-inhibition using Fostamatinib to treat Post-Transplant Immune-mediated Cytopenias).
* Female patients of reproductive potential agree to avoid pregnancy through abstinence or the use two forms of highly effective birth control during and for 1 month after the last study treatment and agree not to donate eggs during this time.
* Male patients of reproductive potential agree to avoid pregnancy of a partner through abstinence or the use two forms of highly effective birth control during and for 1 month after the last study treatment and agree not to donate sperm during this time.

EXCLUSION CRITERIA:

* Severe psychiatric illness or mental deficiency sufficient to make making informed consent impossible
* Positive pregnancy test for women of childbearing age within 1 week or being actively lactating
* Uncontrolled hypertension (systolic blood pressure >140mmHg or diastolic blood pressure >90mmHg)
* ALT or AST >3 times the upper limit of normal
* Patients who have a history of medical disorders, that in the investigator's opinion, could affect the conduct of the study or the absorption, metabolism or excretion of the study drug are excluded.
* Patients with evidence of graft rejection (based on clinical suspicion supported by BM biopsy data and/or chimerism studies and/or MLR)
* Neutropenia, defined as absolute neutrophil count <= 1.0 X 10^9/L
* Non-immune mediated cytopenias. Etiologies including, but not limited to, cytopenias due to HIV infection, lymphoproliferative disorders, myelodysplasia/acute leukemia, drug-induced thrombocytopenia, thrombotic microangiopathies, acute bleeding, consumptive coagulopathy, fever, infections leading to cytopenia, medications induced cytopenias, thrombotic microangiopathies (disseminated intravascular coagulation), splenomegaly or hemophagocytic lymphohistiophagocytosis, relapse of primary disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-11-07 (Actual); Primary Completion 2025-11-07 (Actual); Study Completion 2025-11-07 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects who are able to maintain hematologic recovery | 12 weeks
  Proportion of subjects who are able to maintain hematologic recovery (as defined below) by the end of 12 weeks on the extended access trial (total of 24 weeks fostamatinib treatment). Hematologic recovery is defined as: Hemoglobin >=10 g/dL (or at least >=2 g/dL above baseline) in subjects enrolled with post-transplant anemia. In subjects with symptomatic anemia, a hemoglobin increase of at least >=2 g/dL above baseline is required OR Platelets >= 50 x 109/L (or at least =20 x 10^9/L above baseline) in subjects enrolled with post-transplant thrombocytopenia OR Both of the above criteria in subjects with post-transplant Evan s syndrome

SECONDARY OUTCOMES:
Proportion of subjects who are able to taper off fostamatinib by >33% while maintaining hematologic recovery | 106 weeks
  Hematologic recovery is defined as: Hemoglobin >=10 g/dL (or at least >=2 g/dL above baseline) in subjects enrolled with post-transplant anemia. In subjects with symptomatic anemia, a hemoglobin increase of at least >=2 g/dL above baseline is required OR Platelets >= 50 X 10^9/L (or at least >=20 X 10^9/L above baseline) in subjects enrolled with post-transplant thrombocytopenia OR Both of the above criteria in subjects with post-transplant Evan s syndrome
Change in the dose of other immunosuppressive agents | 12 weeks
  Change in the dose of other immunosuppressive agents in the total 24 weeks on fostamatinib, measured by median daily dose of the immunosuppressant in a week, from week 1 to week 24.
Proportion of subjects who are able to completely taper off fostamatinib while maintaining hematologic recovery | 106 weeks
  Hematologic recovery is defined as: Hemoglobin >=10 g/dL (or at least >=2 g/dL above baseline) in subjects enrolled with post-transplant anemia. In subjects with symptomatic anemia, a hemoglobin increase of at least >=2 g/dL above baseline is required OR Platelets >= 50 X 10^9/L (or at least >=20 X 10^9/L above baseline) in subjects enrolled with post-transplant thrombocytopenia OR Both of the above criteria in subjects with post-transplant Evan s syndrome
Change in corticosteroid dose | 12 weeks
  Change in corticosteroid dose in the total 24 weeks on fostamatinib, measured by median daily weight-based prednisone-equivalent corticosteroid dose from week 1 to week 24.

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Y Hur, D.O., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_000760-H.html